CLINICAL TRIAL: NCT05285644
Title: A Phase 3 Study Evaluating the Safety and Efficacy of AR-15512, a Cold Thermoreceptor Modulator, for the Treatment of Dry Eye Disease (COMET-2)
Brief Title: Study Evaluating the Safety and Efficacy of AR-15512
Acronym: COMET-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR-15512-CS301
Record Dates: First submitted 2022-03-04; First posted 2022-03-17 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.003% AR-15512 (Experimental): 0.003% AR-15512 ophthalmic solution, one drop in each eye twice a day for 90 days
  Interventions: Drug: 0.003% AR-15512 ophthalmic solution
- AR-15512 Vehicle (Placebo Comparator): AR-15512 vehicle ophthalmic solution, one drop in each eye twice a day for 90 days
  Interventions: Drug: AR-15512 vehicle ophthalmic solution

INTERVENTIONS:
Drug: 0.003% AR-15512 ophthalmic solution — Administered via topical ocular instillation
  Arms: 0.003% AR-15512
Drug: AR-15512 vehicle ophthalmic solution — Inactive ingredients administered via topical ocular instillation
  Arms: AR-15512 Vehicle

SUMMARY:
This will be a Phase 3, multicenter, vehicle-controlled, double-masked, randomized study conducted at approximately 20 sites in the United States. All subjects enrolled will have dry eye disease (DED). The study will consist of Screening (Day -14) and Baseline (Day 1) visits as well as visits at Day 7, Day 14, Day 28, and Day 90 (Study Exit) for an individual duration of participation of approximately 15 weeks.

DETAILED DESCRIPTION:
At the end of the Screening Visit, all qualified subjects will be assigned to administer one drop of AR-15512 Vehicle twice a day to both eyes for approximately 14 days (vehicle run-in period). After the vehicle run-in period, subjects will be re-evaluated for signs and symptoms of Dry Eye Disease (DED). Subjects who requalify based on inclusion/exclusion criteria will be enrolled in the study and randomized in a 1:1 ratio to receive 0.003% AR-15512 or AR-15512 Vehicle administered as 1 drop in each eye twice a day for 90 days. At the end of the Day 90 visit, subjects will exit the study.

Aerie Pharmaceuticals was acquired by Alcon on November 22, 2022.

ELIGIBILITY:
Key Inclusion Criteria:

* Signs and symptoms of dry eye disease (DED) at the Screening and Baseline visits;
* Corrected visual acuity of +0.70 logarithm Minimum angle of resolution (LogMAR) or better in both eyes at Screening and Baseline visits;
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* History or presence of any ocular disorder or condition (other than DED) in either eye that would, in the opinion of the investigator, likely interfere with the interpretation of the study results or subject safety;
* Regular use of lid hygiene within 14 days prior to the Screening visit or any planned use during the study;
* Use of artificial tears within 2 hours prior to the Screening visit or anticipated use during the study;
* Medication use as specified in the protocol;
* History or presence of significant systemic disease;
* Other protocol-specified exclusion criteria may apply.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scientific Advisor, Clinical R&D, Study Director — Alcon Research, LLC
Locations (23):
- United States (23):
  - Global Research Management, Inc, Glendale, California
  - Premiere Practice Management, LLC, Torrance, California
  - Vision Institute, Colorado Springs, Colorado
  - The Eye Care Group, Waterbury, Connecticut
  - Segal Drug Trials, Inc., Delray Beach, Florida
  - Michael Washburn Center for Ophthalmic Research, LLC, Indianapolis, Indiana
  - Butchertown Clinical Trials, Louisville, Kentucky
  - Central Maine Eye Care, Lewiston, Maine
  - Moyes Eye Center, Kansas City, Missouri
  - Center for Sight, Henderson, Nevada
  - Core, Inc., Shelby, North Carolina
  - Bergstrom Eye Research, Fargo, North Dakota
  - Verum Research, Eugene, Oregon
  - Erie Retina Research, Erie, Pennsylvania
  - Advancing Vision Research, Goodlettsville, Tennessee
  - Total Eye Care, PA, Memphis, Tennessee
  - Advancing Vision Research, Smyrna, Tennessee
  - Austin Clinical Research, Austin, Texas
  - Valley Retina Institute, PA, Harlingen, Texas
  - Valley Retina Institute, PA, McAllen, Texas
  - Eye Clinics of South Texas, San Antonio, Texas
  - R and R Eye Research, LLC, San Antonio, Texas
  - Alpine Research Organization Inc., Clinton, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pattar GR, Wirta D, Jerkins G, Paauw J, McLaurin EB, Liu A, Evans DG, Kenyon K, Cline N, Gupta PK, Meng I, Senchyna M; COMET-2 and COMET-3 Study Groups. Acoltremon Ophthalmic Solution 0.003% for Signs and Symptoms of Dry Eye Disease: Results of Phase 3 Pivotal COMET-2 and COMET-3 Studies. Ophthalmology. 2025 Sep 30:S0161-6420(25)00605-0. doi: 10.1016/j.ophtha.2025.09.018. Online ahead of print. PMID 41038456

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 23 investigative sites located in the United States.
Pre-assignment Details: This reporting group includes all randomized participants.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Started | 230; 460 eyes | 235; 470 eyes
ITT Population (All randomized subjects) | 230; 460 eyes | 235; 470 eyes
Safety Population (All randomized subjects who have received at least one dose of the investigational product) | 230; 460 eyes | 235; 470 eyes
Completed | 210; 420 eyes | 213; 426 eyes
Not Completed | 20; 40 eyes | 22; 44 eyes
Not completed — Adverse Event | 3 | 3
Not completed — Withdrawal of Consent | 2 | 5
Not completed — Noncompliance | 0 | 4
Not completed — Lost to Follow-up | 4 | 6
Not completed — Disallowed Concurrent Medication | 1 | 1
Not completed — Investigator Decision | 2 | 0
Not completed — Protocol Deviation | 1 | 0
Not completed — As specified in the Clinical Study Report | 7 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle | Total
Number analyzed (Participants) | 230 | 235 | 465
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (13.04) | 59.6 (13.43) | 59.6 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 180 | 353
  Male | 57 | 55 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 34 | 65
  Not Hispanic or Latino | 199 | 201 | 400
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian / Alaska Native | 0 | 1 | 1
  Asian | 24 | 21 | 45
  Black / African American | 35 | 32 | 67
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 168 | 179 | 347
  Multi-racial | 2 | 1 | 3
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 230 | 235 | 465
Unanesthetized Schirmer Test Pre-Drop at Baseline (Day 1) [Mean (Standard Deviation); unit: milllimeter] | 6.2 (5.49) | 5.9 (5.41) | 6.1 (5.45)
Global SANDE Score at Baseline (Day 1) [Mean (Standard Deviation); unit: millimeter] | 72.7 (12.16) | 72.7 (11.74) | 72.7 (11.94)
SANDE Frequency Score at Baseline (Day 1) [Mean (Standard Deviation); unit: millimeter] | 75.2 (13.77) | 75.0 (13.74) | 75.1 (13.74)
SANDE Severity Score at Baseline (Day 1) [Mean (Standard Deviation); unit: millimeter] | 71.1 (13.28) | 71.3 (12.64) | 71.2 (12.95)
Eye Dryness Score at Baseline (Day 1) [Mean (Standard Deviation); unit: millimeter] | 72.8 (14.77) | 71.5 (13.54) | 72.2 (14.16)
Ocular Discomfort Score at Baseline (Day 1) [Mean (Standard Deviation); unit: millimeter] | 74.4 (12.67) | 73.4 (12.11) | 73.9 (12.39)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Achieved Equal to or Greater Than 10 Millimeter Increase From Pre-drop at Baseline to Post-drop on Day 14 in Study Eye Unanesthetized Schirmer Score
Description: The Schirmer test measures tear production using a filter paper placed on the lower eyelid. The amount of wetting was recorded on a scale from 0 millimeters (mm) (no tear production) to 35 mm (maximum). The test was performed at Day 1 prior to drop exposure and at Day 14 following drop exposure. An increased score represents a positive outcome. One eye (study eye) contributed data to the analysis.
Time Frame: Baseline (Day 1) pre-drop; Day 14 post-drop
Population: ITT population comprising all randomized subjects. This analysis uses multiple imputation methodology.
Measure: Number; unit: percentage of subjects
Units Other Than Participants: eyes
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 230 | 235
Number analyzed (eyes) | 230 | 235
percentage of subjects | 42.6 | 8.2
Statistical Analysis 1: Comparison: 0.003% AR-15512 vs AR-15512 Vehicle; The primary estimand targeted the treatment effect attributable to the randomly assigned treatment, regardless of compliance to study treatment and assuming subjects who discontinued due to lack of efficacy, AEs, or disallowed concurrent treatments followed the behavior of subjects in the reference arm for the duration of the study and subjects who discontinued for other reasons would have followed the behavior of subjects who were still in the study under same randomly assigned treatment; Test type: Other — Difference (2-sided); p < 0.0001, Pearson's Chi-squared test — Multiple imputation methodology was implemented in handling missing data, both related to and unrelated to intercurrent events; Difference in Percentages = 34.4, 95% CI 2-sided [26.9 to 42.0] — Difference equals 0.003% AR-15512 minus AR-15512 Vehicle; For binary endpoint, the underlying continuous measurement of unanesthetized Schirmer score was imputed, change score calculated and then dichotomized to ascertain attainment of greater than or equal to 10 millimeter increase from pre-drop baseline

2. Secondary Outcome: Least Squares Mean Change From Baseline in Global Symptom Assessment iN Dry Eye (SANDE) Score on Day 28
Description: The SANDE questionnaire assesses the frequency and severity of symptoms using 2 unique, 100 mm Visual Analog Scales to mark the frequency (0=rarely, 100=all the time) and severity (0=very mild, 100=very severe) of dry eye symptoms (prior to drop exposure). The 2 scores were multiplied and a square root was obtained for a resultant overall Global SANDE score of 0 to 100 where 0 represents no symptoms and 100 is maximum symptoms. A negative change indicates a better outcome. This was a subject based assessment (single score for both eyes).
Time Frame: Baseline (Day 1); Day 28
Population: ITT population comprising all randomized subjects. This analysis uses multiple imputation methodology.
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 230 | 235
millimeter | -19.7 (1.61) | -14.7 (1.58)
Statistical Analysis 1: Comparison: 0.003% AR-15512 vs AR-15512 Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Other — Difference (2-sided); p = 0.0138, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; Least Squares Mean Difference = -5.1, 95% CI 2-sided [-9.1 to -1.0], Standard Error of Mean 2.06 — Difference equals 0.003% AR-15512 minus AR-15512 Vehicle

3. Secondary Outcome: Least Squares Mean Change From Pre-drop Baseline in Unanesthetized Schirmer Score on Post-drop Day 14 (Study Eye)
Description: The Schirmer test measures tear production using a filter paper placed on the lower eyelid. The amount of wetting was recorded on a scale from 0 millimeters (mm) (no tear production) to 35 mm (maximum). The test was performed at Day 1 prior to drop exposure and at Day 14 following drop exposure. The Day 14 value was compared to the Day 1 value. A positive change indicates a better outcome. One eye (study eye) contributed data to the analysis.
Time Frame: Baseline (Day 1) pre-drop; Day 14 post-drop
Population: ITT population comprising all randomized subjects. This analysis uses multiple imputation methodology.
Measure: Least Squares Mean (Standard Error); unit: millimeter
Units Other Than Participants: eyes
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 230 | 235
Number analyzed (eyes) | 230 | 235
millimeter | 9.8 (0.55) | 2.6 (0.54)
Statistical Analysis 1: Comparison: 0.003% AR-15512 vs AR-15512 Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Other — Difference (2-sided); p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; Least Squares Mean Difference = 7.2, 95% CI 2-sided [5.8 to 8.6], Standard Error of Mean 0.70; Difference equals 0.003% AR-15512 minus AR-15512 Vehicle

4. Secondary Outcome: Percentage of Subjects Who Achieved Equal to or Greater Than 10 Millimeter Increase From Pre-drop at Baseline to Post-drop on Day 1 in Study Eye Unanesthetized Schirmer Score
Description: The Schirmer test measures tear production using a filter paper placed on the lower eyelid. The amount of wetting was recorded on a scale from 0 millimeters (mm) (no tear production) to 35 mm (maximum). The test was performed at Day 1 prior to drop exposure and at Day 1 following drop exposure. The Day 1 post-drop score was compared to the Day 1 pre-drop score. An increased score represents a positive outcome. One eye (study eye) contributed data to the analysis.
Time Frame: Baseline (Day 1) pre-drop; Day 1 post-drop
Population: ITT population comprising all randomized subjects. This analysis uses multiple imputation methodology.
Measure: Number; unit: percentage of subjects
Units Other Than Participants: eyes
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 230 | 235
Number analyzed (eyes) | 230 | 235
percentage of subjects | 36.1 | 9.4
Statistical Analysis 1: Comparison: 0.003% AR-15512 vs AR-15512 Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Other — Difference (2-sided); p < 0.0001, Pearson's Chi-squared test — [p-value comment as in outcome 1, analysis 1]; Difference in Percentages = 26.7, 95% CI 2-sided [19.5 to 34.0] — Difference equals 0.003% AR-15512 minus AR-15512 Vehicle; [other analysis details as in outcome 1, analysis 1]

5. Secondary Outcome: Least Squares Mean Change From Pre-drop Baseline in Unanesthetized Schirmer Score on Post-drop Day 1 (Study Eye)
Description: The Schirmer test measures tear production using a filter paper placed on the lower eyelid. The amount of wetting was recorded on a scale from 0 millimeters (mm) (no tear production) to 35 mm (maximum). The test was performed at Day 1 prior to drop exposure and at Day 1 following drop exposure. The Day 1 post-drop score was compared to the Day 1 pre-drop score. A positive change over time indicates a better outcome. One eye (study eye) contributed data to the analysis.
Time Frame: Baseline (Day 1) pre-drop; Day 1 post-drop
Population: ITT population comprising all randomized subjects. This analysis uses multiple imputation methodology.
Measure: Least Squares Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: eyes
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 230 | 235
Number analyzed (eyes) | 230 | 235
millimeter | 8.9 (0.53) | 2.7 (0.52)
Statistical Analysis 1: Comparison: 0.003% AR-15512 vs AR-15512 Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Other — Difference (2-sided); p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; Least Squares Mean Difference = 6.2, 95% CI 2-sided [4.9 to 7.5], Standard Error of Mean 0.68 — Difference equals 0.003% AR-15512 minus AR-15512 Vehicle

6. Secondary Outcome: Percentage of Subjects Who Achieved Equal to or Greater Than 10 Millimeter Increase From Pre-drop at Baseline to Post-drop on Day 90 in Study Eye Unanesthetized Schirmer Score
Description: The Schirmer test measures tear production using a filter paper placed on the lower eyelid. The amount of wetting was recorded on a scale from 0 millimeters (mm) (no tear production) to 35 mm (maximum). The test was performed at Day 1 prior to drop exposure and at Day 90 following drop exposure. The Day 90 post-drop score was compared to the Day 1 pre-drop score. An increased score represents a positive outcome. One eye (study eye) contributed data to the analysis.
Time Frame: Baseline (Day 1) pre-drop; Day 90 post-drop
Population: ITT population comprising all randomized subjects. This analysis uses multiple imputation methodology.
Measure: Number; unit: percentage of subjects
Units Other Than Participants: eyes
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 230 | 235
Number analyzed (eyes) | 230 | 235
percentage of subjects | 46.7 | 13.6
Statistical Analysis 1: Comparison: 0.003% AR-15512 vs AR-15512 Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Other — Difference (2 sided); p < 0.0001, Pearson's Chi-squared test — [p-value comment as in outcome 1, analysis 1]; Difference in Percentages = 33.1, 95% CI 2-sided [24.8 to 41.4] — Difference equals 0.003% AR-15512 minus AR-15512 Vehicle; [other analysis details as in outcome 1, analysis 1]

7. Secondary Outcome: Least Squares Mean Change From Pre-drop Baseline in Unanesthetized Schirmer Score on Post-drop Day 90 (Study Eye)
Description: The Schirmer test measures tear production using a filter paper placed on the lower eyelid. The amount of wetting was recorded on a scale from 0 millimeters (mm) (no tear production) to 35 mm (maximum). The test was performed at Day 1 prior to drop exposure and at Day 90 following drop exposure. The Day 90 post-drop score was compared to the Day 1 pre-drop score. A positive change over time indicates a better outcome. One eye (study eye) contributed data to the analysis.
Time Frame: Baseline (Day 1) pre-drop; Day 90 post-drop
Population: ITT population comprising all randomized subjects. This analysis uses multiple imputation methodology.
Measure: Least Squares Mean (Standard Error); unit: millimeter
Units Other Than Participants: eyes
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 230 | 235
Number analyzed (eyes) | 230 | 235
millimeter | 10.7 (0.59) | 3.1 (0.57)
Statistical Analysis 1: Comparison: 0.003% AR-15512 vs AR-15512 Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Other — Difference (2-sided); p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; Least Squares Mean Difference = 7.5, 95% CI 2-sided [6.0 to 9.0], Standard Error of Mean 0.76 — Difference equals 0.003% AR-15512 minus AR-15512 Vehicle

8. Secondary Outcome: Least Squares Mean Change From Baseline in Global SANDE Score on Day 90
Description: as for outcome 2
Time Frame: Baseline (Day 1); Day 90
Population: ITT population comprising all randomized subjects. This analysis uses multiple imputation methodology.
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 230 | 235
millimeter | -23.5 (1.78) | -20.7 (1.77)
Statistical Analysis 1: Comparison: 0.003% AR-15512 vs AR-15512 Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Other — Difference (2-sided); p = 0.2184, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; Least Squares Mean Difference = -2.8, 95% CI 2-sided [-7.3 to 1.7], Standard Error of Mean 2.28 — Difference equals 0.003% AR-15512 minus AR-15512 Vehicle

9. Secondary Outcome: Least Squares Mean Change From Baseline in SANDE Frequency Score on Day 90
Description: The SANDE questionnaire assesses the frequency of dry eye disease symptoms. Subjects used a 100 mm Visual Analog Scale (VAS) to mark the frequency of symptoms where 0=rarely and 100=all the time. A higher SANDE frequency score indicates greater symptoms of dryness and/or irritation. The questionnaire was completed at Day 1 and Day 90 prior to drop exposure (both visits). The Day 90 value was compared to the Day 1 value. A negative change indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1); Day 90
Population: ITT population comprising all randomized subjects. This analysis uses multiple imputation methodology.
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 230 | 235
millimeter | -22.8 (1.89) | -20.1 (1.89)
Statistical Analysis 1: Comparison: 0.003% AR-15512 vs AR-15512 Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Other — Difference (2-sided); p = 0.2660, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; Least Squares Mean Difference = -2.7, 94% CI 2-sided [-7.5 to 2.1], Standard Error of Mean 2.43 — Difference equals 0.003% AR-15512 minus AR-15512 Vehicle

10. Secondary Outcome: Least Squares Mean Change From Baseline in SANDE Severity Score on Day 90
Description: The SANDE questionnaire assesses the severity of dry eye disease symptoms. Subjects used a 100 mm Visual Analog Scale (VAS) to mark the severity of symptoms where 0=very mild and 100=very severe. A higher SANDE severity score indicates greater symptoms of dryness and/or irritation. The questionnaire was completed at Day 1 and Day 90 prior to drop exposure (both visits). The Day 90 value was compared to the Day 1 value. A negative change indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1); Day 90
Population: ITT population comprising all randomized subjects. This analysis uses multiple imputation methodology.
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 230 | 235
millimeter | -23.1 (1.87) | -20.5 (1.84)
Statistical Analysis 1: Comparison: 0.003% AR-15512 vs AR-15512 Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Other — Difference (2-sided); p = 0.2741, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; Least Squares Mean Difference = -2.6, 95% CI 2-sided [-7.2 to 2.0], Standard Error of Mean 2.37 — Difference equals 0.003% AR-15512 minus AR-15512 Vehicle

11. Secondary Outcome: Least Squares Mean Change From Baseline in Eye Dryness Score (EDS) on Day 90
Description: The subject used a 100 mm Visual Analog Scale (VAS) to mark their eye dryness, where 0=no eye dryness and 100=maximum eye dryness. Eye dryness was assessed at Day 1 and Day 90 prior to drop exposure (both visits). A higher eye dryness score indicates greater dryness. The Day 90 value was compared to the Day 1 value. A negative change indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1); Day 90
Population: ITT population comprising all randomized subjects. This analysis uses multiple imputation methodology.
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 230 | 235
millimeter | -22.5 (1.89) | -19.1 (1.84)
Statistical Analysis 1: Comparison: 0.003% AR-15512 vs AR-15512 Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Other — Difference (2-sided); p = 0.1590, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; Least Squares Mean Difference = -3.4, 95% CI 2-sided [-8.2 to 1.3], Standard Error of Mean 2.43 — Difference equals 0.003% AR-15512 minus AR-15512 Vehicle

12. Secondary Outcome: Least Squares Mean Change From Baseline in Ocular Discomfort Score (ODS) on Day 90
Description: The subject used a 100 mm Visual Analog Scale (VAS) to mark their eye dryness, where 0=no ocular discomfort and 100 mm=maximum ocular discomfort. A higher ocular discomfort score indicates greater discomfort. Ocular discomfort was assessed at Day 1 and Day 90 prior to drop exposure (both visits). The Day 90 value was compared to the Day 1 value. A negative change indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1); Day 90
Population: ITT population comprising all randomized subjects. This analysis uses multiple imputation methodology.
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 230 | 235
millimeter | -32.2 (2.06) | -28.2 (2.04)
Statistical Analysis 1: Comparison: 0.003% AR-15512 vs AR-15512 Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Other — Difference (2-sided); p = 0.1369, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-9.2 to 1.3], Standard Error of Mean 2.67 — Difference equals 0.003% AR-15512 minus AR-15512 Vehicle

ADVERSE EVENTS:
Time Frame: An adverse event was (AE) defined as any untoward medical occurrence associated with the administration of the drug in humans, whether or not considered drug related. AE's were collected from time of consent until study exit, approximately 15 weeks. The safety population includes all randomized subjects who have received at least one dose of the investigational product. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator.
Description: All participants were monitored for serious and other ocular and nonocular AEs. All-Cause Mortality was not monitored for the ocular arms. However, the nonocular AE arms were not considered at Risk for ocular adverse event terms as the arms are reporting nonocular-specific AEs. Similarly, the ocular AE arms were not considered at Risk for nonocular adverse event terms as the arms are reporting ocular-specific AEs.
Groups:
- Pretreatment: AEs reported in this group occurred prior to treatment with the study drug and include the 2-week vehicle run-in.
- 0.003% AR-15512 Ocular; 0.003% AR-15512 Nonocular: AEs reported in this group occurred during the 0.003% AR-15512 ophthalmic solution treatment period.
- AR-15512 Vehicle Ocular; AR-15512 Vehicle Nonocular: AEs reported in this group occurred during the AR-15512 vehicle ophthalmic solution treatment period.
Arm/Group | Pretreatment | 0.003% AR-15512 Ocular | 0.003% AR-15512 Nonocular | AR-15512 Vehicle Ocular | AR-15512 Vehicle Nonocular
All-Cause Mortality (participants affected / at risk) | 0/465 | 0/0 | 0/230 | 0/0 | 0/235
Serious Adverse Events (participants affected / at risk) | 1/465 | 0/230 | 1/230 | 0/235 | 6/235
Other Adverse Events (participants affected / at risk) | 4/465 | 120/230 | 0/230 | 10/235 | 0/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pretreatment (N=465) | 0.003% AR-15512 Ocular (N=230) | 0.003% AR-15512 Nonocular (N=230) | AR-15512 Vehicle Ocular (N=235) | AR-15512 Vehicle Nonocular (N=235)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0/0 (0) | 0 (0) | 0/0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0/0 (0) | 0 (0) | 0/0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0/0 (0) | 0 (0) | 0/0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0/0 (0) | 0 (0) | 0/0 (0) | 1 (1)
Norovirus infection (Infections and infestations) | 0 (0) | 0/0 (0) | 0 (0) | 0/0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0/0 (0) | 0 (0) | 0/0 (0) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0/0 (0) | 1 (1) | 0/0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0/0 (0) | 0 (0) | 0/0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0/0 (0) | 0 (0) | 0/0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0/0 (0) | 0 (0) | 0/0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0/0 (0) | 0 (0) | 0/0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pretreatment (N=465) | 0.003% AR-15512 Ocular (N=230) | 0.003% AR-15512 Nonocular (N=230) | AR-15512 Vehicle Ocular (N=235) | AR-15512 Vehicle Nonocular (N=235)
Instillation site pain (General disorders) | 4 (4) | 120 (125) | 0/0 (0) | 10 (10) | 0/0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/44/NCT05285644/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT05285644/SAP_001.pdf